CLINICAL TRIAL: NCT01021423
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-Controlled, First Line Maintenance Study Of Lenalidomide (Revlimid®) In Patients With Mantle-Cell Lymphoma
Brief Title: A Study to Evaluate the Efficacy of Lenalidomide as Maintenance Therapy After Completion of First-line Combination Chemotherapy in Patients With Mantle Cell Lymphoma (MCL).
Acronym: RENEW
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by sponsor due to new unpublished data that rendered the current design of the study no longer clinically relevant. There were no safety concerns.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-MCL-003
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma; CC-5013; Revlimid; Lenalidomide
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide - 15 mg orally once daily on Days 1-21 of every 28-day cycle for a maximum of 2 years or until disease progression, unacceptable toxicity develops or voluntary withdrawal.
  Interventions: Drug: Lenalidomide
- Placebo (Experimental): Placebo (identical matched capsule) orally once daily on Days 1-21 of every 28-day cycle for a maximum of 2 years or until disease progression, unacceptable toxicity develops or voluntary withdrawal.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lenalidomide — 15 mg orally once daily on Days 1-21 of every 28-day cycle for a maximum of 2 years or until disease progression, unacceptable toxicity develops or voluntary withdrawal.
  Other Names: Revlimid
  Arms: Lenalidomide
Other: Placebo — Placebo (identical matched capsule) orally once daily on Days 1-21 of every 28-day cycle for a maximum of 2 years or until disease progression, unacceptable toxicity develops or voluntary withdrawal.
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy of lenalidomide as maintenance therapy after completion of first-line combination chemotherapy in patients with mantle cell lymphoma (MCL) who are not candidates for transplantation and have achieved partial response (PR) or complete response (CR).

This study was prematurely terminated by the sponsor in light of new unpublished data that rendered the current design of the study no longer clinically relevant. A study design with the control arm of no active treatment was no longer appropriate. The termination of the trial was not based on any safety concerns in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven mantle cell non-Hodgkin's lymphoma,
* One of the following first-line induction chemotherapy regimens with rituximab: (1) combination regimen containing all of the following components: cyclophosphamide, vincristine, adriamycin and a glucocorticoid; (2) Fludarabine containing regimen such as FC (fludarabine, cyclophosphamide)
* Achieved a PR or better response after the first-line induction chemotherapy regimen (assessed by 2007 Revised Response Criteria for Malignant Lymphoma)
* ECOG performance status score of ≤ 2
* Willing to follow pregnancy precaution

Exclusion Criteria:

* Patients who have received more than 1 line of induction chemotherapy;
* Patients who have received less than 4 cycles of R-CHOP, R-CHOP-like, or R-FC are ineligible;
* Patients who achieved stable disease or progressive disease as best response with first line-induction chemotherapy;
* Any of the following laboratory abnormalities:
* Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5*10^9/L)
* Platelet count < 60,000/mm^3 (60*10^9/L)
* Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT)) > 3.0 times upper limit of normal (ULN), except in patients with documented liver involvement by lymphoma
* Serum bilirubin > 1.5 times ULN, except in case of Gilbert's Syndrome and documented liver involvement by lymphoma
* Calculated creatinine clearance (i.e. Cockcroft-Gault formula) of < 30 mL /min
* Active or any history of central nervous system (CNS) lymphoma or leptomeningeal involvement by lymphoma
* Subjects at high risk for deep vein thrombosis (DVT) not willing to take DVT prophylaxis
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dreyling, Prof. Dr, Principal Investigator — Medizinische Klinik III der Universität München
Locations (92):
- United States (13):
  - Sharp Healthcare Oncology Associates of San Diego, San Diego, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Providence Cancer Center, Indianapolis, Indiana
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Arena Oncology Associates, Lake Success, New York
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Virginia Health Systems, Charlottesville, Virginia
- Czechia (5):
  - Fakultni nemocnice Hradec Králové II. Interni klinika-Oddeleni klinicke hematologie, Hradec Králové
  - Fakultni Nemocnice Olomouc, Hemato-Onkologicka Klinika, Olomouc
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice, Prague
  - Clinic of Oncology Faculty Hospital Motol, Prague
- France (19):
  - CHU Amiens Sud, Centre de Recherche Clinique - Pharmacologie Clinique, Amiens
  - CHU Hôpital Hotel Dieu, Angers
  - CHU ESTAING, Service d'Hématologie, Clermont-Ferrand
  - Hôpital Henri Mondor Unité Hémopathies Lymphoides, Créteil
  - CHD Les Oudairies, Service d'Oncologie Hématologie, La Roche-sur-Yon
  - Centre Hospitalier Lyon Sud, Pavillon Marcel Bérard 1F Hématologie, La Tronche
  - CHRU - Hôpital Claude Huriez, Lille
  - CHU Montpellier - Hôpital Saint Eloi Hématologie et Oncologie Médicale, Montpellier
  - CHRU - Hotel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - CHRU - Hôpital du Haut Lévêque, maladies du sang, Centre François Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pavillon Marcel Bérard 1F Hématologie, Pierre-Bénite
  - CHU de Poitiers, Pôle Régional de Cancérologie, Service d'Oncologie Hématologie et Thérapie Cellulaire, Poitiers
  - CHU de Reims, Hôpital Robert Debré, Hématologie Clinique, Reims
  - Hôpital Pontchaillou Hématologie Clinique, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital Purpan CHU de Toulouse, Toulouse
  - Hôpital Bretonneau - CHU Tours, Tours
  - CHU de Nancy Hôpital de Brabois, Service d'Hématologie et Médecine Interne, Vandœuvre-lès-Nancy
- Germany (7):
  - Universitätsklinikum Essen Zentrum für Innere Medizin, Essen
  - Universitätsklinikum Freiburg - Medizinische Klinik - Abteilung Innere Medizin I: Hämatologie und Onkologie, Freiburg im Breisgau
  - UKG Universitätsklinikum Göttingen Zentrum Innere Medizin Hämatologie / Onkologie, Göttingen
  - Asklepios Klinik St. Georg - Abteilung für Hämatologie und Stammzelltransplantation, Hamburg
  - Städtisches Klinikum Karlsruhe - Hämatologie / Onkologie Karlsruhe, Karlsruhe
  - Klinikum der Universität München - Großhadern, Medizinische Klinik III, München
  - Universitaetsklinikum Tuebingen, Tübingen
- Israel (2):
  - Soroka Medical Center The Institute of Hematology, Beersheba
  - Davidoff Cancer Center The Institute of Hematology, Petah Tikva
- Italy (16):
  - Az. Osp. SS.Antonio e Biagio SC Ematologia, Alessandria
  - Ospedale Regionale di Bolzano - Divisione di Ematologia, Bolzano
  - Hematology Dept, Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria "San Martino", Genova
  - Az. Osp. Ospedali Riuniti Papardo - Piemonte - S.C. Ematologia, Messina
  - A,O Ospedale Niguarda Ca Granda Dept Hematology, Milan
  - Fondazione San Raffaele del Monte Tabor I.R.C.C.S., Milan
  - Istituto Nazionale Tumori Fondazione "G. Pascale" - Oncoematologia, Napoli
  - Università del Piemonte Orientale "Amedeo Avogadro", Novara
  - Policlinico San Matteo - Dip. Di Ematologia, Pavia
  - Az. Osp. Bianchi Melacrino Morelli, Div. Di Ematologia, Reggio Calabria
  - Università Cattolica del Sacro Cuore Policlinico A. Gemelli, Roma
  - IRCCS Casa Sollievo della Sofferenza Div. Di Oncoematologia, S.Giovanni Rotondo (FG)
  - Azienda Sanitaria Ospedaliera San Giovanni Battista (Molinette), Torino
  - Ospedale Cardinale G. Panico - Ematologia e Immunoematologia, Tricase
  - Clinica Ematologica - DIRM Azienda Ospedaliera Universitaria, Udine
- Poland (3):
  - Małopolskie Centrum Medyczne, Krakow
  - Wojewodzki Szpital Specjalistczny im. Mikolaja Kopernika, Lodz
  - Dolnoslaskie Centrum Transplantacji Komórkowych, Wroclaw
- Portugal (3):
  - Serviço de Hematologia, Coimbra
  - Instituto Português de Oncologia (IPO) de Lisboa, Lisbon
  - Instituto Português de Oncologia (IPO) do Porto, Porto
- Centro de Cancer, Hospital Espanol Auxilio de Puerto Rico, San Juan, Puerto Rico
- Russia (8):
  - Republican Clinical Oncological Dispensary, Kazan'
  - Russian Oncological Research Centre, Moscow
  - Perm Regional Clinical Hospital, Perm
  - Russian Scientific-research Institute of Hematology and Transfusiology of Federal Medical-biological agency, Saint Petersburg
  - State Educational Institution of High Professional Education, Saint Petersburg
  - Federal Center of Heart, Blood and Endocrinology n.a. V.A. Almazov Rosmedtechnologies, Saint Petersburg
  - State Healthcare Institution "Volgograd Regional Clinical OncologyDispensary #1, Volgograd
  - Sverdlovsk Regional Clinical Hospital - Volgogradskaya, Yekaterinburg
- Spain (7):
  - Hospital Universitario Vall d´Hebrón Hematology Department, Barcelona
  - Hospital de Madrid Norte- Sanchinarro, Madrid
  - Hospital Costa del Sol, Oncology, Marbella (Málaga)
  - C. H. de Orense, Ourense
  - Clinica Universitaria de Navarra, Hematology, Pamplona
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Marques de Valdecilla, Santander
- United Kingdom (8):
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Torbay Hospital, County of Devon
  - Royal Devon & Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts & The London NHS Trust Medical Oncology, London
  - Derriford Hospital, Plymouth
  - Salisbury NHS Foundation Trust, Haematology, Salisbury
  - St Helens Hospital, Lilac Lower Ground, St Helens

REFERENCES:
- [Derived] Vose JM, Habermann TM, Czuczman MS, Zinzani PL, Reeder CB, Tuscano JM, Lossos IS, Li J, Pietronigro D, Witzig TE. Single-agent lenalidomide is active in patients with relapsed or refractory aggressive non-Hodgkin lymphoma who received prior stem cell transplantation. Br J Haematol. 2013 Sep;162(5):639-47. doi: 10.1111/bjh.12449. Epub 2013 Jul 9. PMID 23834234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified according to 1) the type of first-line induction chemotherapy (anthracycline-based, fludarabine-based, or rituximab-bendamustine combination therapy) and 2) the response to first-line induction chemotherapy (complete response or partial response).
Period: Overall Study
Arm/Group | Lenalidomide | Placebo
Started | 4 (One participant discontinued treatment (continued in the study) due to an AE) | 5 (One participant discontinued treatment (continued in the study) due to disease progression)
Completed | 0 | 0
Not Completed | 4 | 5
Not completed — Study terminated | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (4.65) | 73.0 (6.89) | 75.1 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Category 0 = Fully active, able to carry on all pre-diseases performance without restriction; Category 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g. light housework, office work).
  participants
    Status = 0 | 4 | 3 | 7
    Status = 1 | 0 | 2 | 2
Response of Mantle Cell Lymphoma (MCL) to chemotherapy at enrollment [Number; unit: participants] — Participants' response to first-line chemotherapy. Response evaluation was as defined by 2007 Revised Response Criteria for Malignant Lymphoma (Cheson 2007). Complete response (CR) is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms if present before therapy. Partial response (PR) is defined as the regression of measurable disease and no appearance of new sites of disease. For full definitions, please refer to the 2007 Revised Response Criteria for Malignant Lymphoma (Cheson 2007).
  participants
    Complete response | 3 | 1 | 4
    Partial response | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization into the study to the first observation of disease progression or death due to any cause. Progression, as defined by the 2007 Revised Response Criteria for Malignant Lymphoma (Cheson, 2007), is any new lesion or increase by 50% of previously involved sites from nadir.
  Study terminated prematurely. Analysis not conducted.
Time Frame: up to 7 years
Population: Study terminated prematurely. Analysis not performed.
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death from any cause.
  Study terminated prematurely. Analysis not conducted.
Time Frame: up to 7 years
Population: Study terminated prematurely. Analysis not performed.
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Participants with treatment-emergent adverse events (TEAEs) during the treatment period plus 30 days. A participant with multiple occurrences of an adverse event within a category is counted only once in that category. Adverse events were evaluated by the investigator.
  The National Cancer Institute (NCI)'s Common Toxicity Criteria for AEs (NCI CTC) was used to grade AE severity. Severity grade 3= severe and undesirable AE. Severity grade 4= life-threatening or disabling AE.
Time Frame: up to 9 months
Population: Safety population of participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 4 | 5
participants
  At least one TEAE | 4 | 4
  At least one TEAE related to study drug | 3 | 2
  At least one NCI CTC grade 3-4 TEAE | 1 | 1
  At least one NCI CTC grade 3-4 related to drug | 1 | 1
  At least one serious TEAE | 1 | 0
  At least one serious TEAE related to drug | 1 | 0
  TEAE leading to discontinuation of drug | 1 | 0
  Related TEAE leading to discontinuation of drug | 1 | 0
  TEAE leading to dose reduction or interruption | 1 | 1
  Related TEAE - dose reduction or interruption | 1 | 1

4. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from the date of randomization until the first date of documented disease progression.
  Study terminated prematurely. Analysis not conducted.
Time Frame: up to 7 years
Population: Study terminated prematurely. Analysis not conducted.
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from randomization until the date at which a participant was removed from treatment due to progression, toxicity, refusal or death or received another Non-Hodgkin Lymphoma (NHL) therapy, whichever occurs first.
Time Frame: up to 2 years
Population: Study terminated prematurely. Analysis not conducted.
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Participants With a Tumor Response
Description: Number of participants with a measurable tumor at time of randomization who achieve a response. Complete response (CR) is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms if present before therapy. Partial response (PR) is defined as the regression of measurable disease and no appearance of new sites of disease. For full definitions, please refer to the 2007 Revised Response Criteria for Malignant Lymphoma (Cheson 2007).
  Study terminated prematurely. Analysis not conducted.
Time Frame: up to 7 years
Population: Study terminated prematurely. Analysis not conducted.
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events occurred during the treatment period, plus 30 days. Due to early termination, the longest experience was 245 days.
Arm/Group | Lenalidomide | Placebo
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=4) | Placebo (N=5)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=4) | Placebo (N=5)
Herpes zoster (Infections and infestations) | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Viral rash (Infections and infestations) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Asthemia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Libido decrease (Psychiatric disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study terminated early. Most analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, agreement to be established before publication.
* Multicenter publication has priority over subset (single center) publication, for duration of 1 year after study completion.
* Individual investigators have publication right after multicenter publication is complete or 1 year after study completion, whichever is first. Celgene has the right to comment and right to ask delay of publication for up to 90 days.